CLINICAL TRIAL: NCT07254650
Title: A Phase IIb, Randomized, Double-Blinded, Three-Arm Clinical Trial: The Study of Liposomal Bupivacaine Via Intercostal Nerve Block, Serratus Anterior Plane Block, or Combination Block for Pain Control After Robotic Thoracic Surgery
Brief Title: Combination Versus Alone Liposomal Bupivacaine Blocks in Minimally Invasive Thoracic Surgery-1
Acronym: CALMS-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The University of Texas at Dallas (Other); Simmons Cancer Center (Other)
Responsible Party: Principal Investigator, Inderpal Sarkaria, Chief of the Division of Thoracic Surgery and Professor of Thoracic Surgery at University of Texas Southwestern Medical Center, and Robert Tucker Hayes Foundation Distinguished Chair in Cardiothoracic Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2025-1629
Record Dates: First submitted 2025-11-04; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: Exparel®; Liposomal Bupivacaine; Multi-Level Intercostal Nerve Block; Serratus Anterior Plane Block; Robotic-Assisted Thoracic Surgery; Adult; Pulmonary Wedge Resection; Lobectomy; Pulmonary Segmentectomy; Pneumonectomy; Minimally-Invasive Thoracic Surgery; Pain Control; Regional Anesthetic Block
MeSH Terms: conditions — Lung Neoplasms; Disease; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: The 3 treatment arms are as follows for intra-operative injection of Liposomal Bupivacaine (LipoB) as a regional anesthetic block:
  * Arm 1: Entire dose (20mL) of LipoB and (20mL) Marcaine® injected locally via multi-level intercostal nerve block (ICNB)
  * Arm 2: Entire dose (20mL) of LipoB and (20mL) Marcaine® injected regionally as serratus anterior plane block (SAPB)
  * Arm 3: Half dose (10mL) of LipoB and (10mL) Marcaine® mixed with 20cc saline injected as ICNB, half dose (10mL) of LipoB and (10mL) Marcaine® mixed with 20cc saline injected as SAPB.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and outcomes-assessors (floor or ICU nurses, research nurses, any person administering study questionnaires) will be blinded. Provider administering regional block (surgeon or anesthesiologist) will not be blinded but will not collect post-operative outcomes data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 "LipoB-I": Liposomal Bupivacaine via Multi-Level Intercostal Nerve Block (Experimental): Patients randomized to Arm 1 "LipoB-I" will receive Liposomal Bupivacaine (LipoB) as an intra-operative multi-level intercostal nerve block containing 266mg (20mL) of Liposomal Bupivacaine (Exparel®) combined with 50mg (20mL) of 0.25% Bupivacaine Hydrochloride, for a total of 40mL for the block.
  Interventions: Procedure: Arm 1 "LipoB-I": Liposomal Bupivacaine via Multi-Level Intercostal Nerve Block
- Arm 2 "LipoB-S": Liposomal Bupivacaine via Serratus Anterior Plane Block (Experimental): Patients randomized to Arm 2 "LipoB-S" will receive Liposomal Bupivacaine (LipoB) as an intra-operative serratus anterior plane block containing 266mg (20mL) of Liposomal Bupivacaine (Exparel®) combined with 50mg (20mL) of 0.25% Bupivacaine Hydrochloride, for a total of 40mL for the block.
  Interventions: Procedure: Arm 2 "LipoB-S": Liposomal Bupivacaine via Serratus Anterior Plane Block
- Arm 3 "LipoB-C": Liposomal Bupivacaine via Combination Block (Experimental): Patients randomized to Arm 3 "LipoB-C" will receive Liposomal Bupivacaine (LipoB) as an intra-operative combination block (multi-level intercostal nerve block [ICNB] and serratus anterior plane block [SAPB]) with half the dose of Liposomal Bupivacaine administered in each block. Block solutions are as follows:
  10mL LipoB mixed with 10mL 0.25% Bupivacaine Hydrochloride and 20mL of saline, administered as SAPB by anesthesiologist immediately prior to incision while in the operating room
  AND
  10mL LipoB mixed with 10mL 0.25% Bupivacaine Hydrochloride and 20mL of saline administered as ICNB prior to closure in at least 5 intercostal spaces as determined by administering surgeon while in the operating room.
  Interventions: Procedure: Arm 3 "LipoB-C": Liposomal Bupivacaine Administered via Combination Block

INTERVENTIONS:
Procedure: Arm 1 "LipoB-I": Liposomal Bupivacaine via Multi-Level Intercostal Nerve Block — The anesthetic mixture is prepared by combining 266 mg (20 mL) of Liposomal Bupivacaine (Exparel®) with 50 mg (20 mL) of 0.25% Bupivacaine Hydrochloride, creating a mixture of 40 mL. This mixture is administered via multi-level intercostal nerve block (ICNB).
  One injection is administered by a surgeon per intercostal space (ICS), given at the origin of the nerve space junction where the nerve and the inferior aspect of the rib meet after the nerve immerges from the intervertebral foramina. At least 5 mL, and no more than 8mL, will be injected in each ICS with the ideal injection consisting of 3 mL just beneath the pleura and 5 mL deeper in the intercostal muscular tissue for a total of 8 mL per ICS. Injections will be completed utilizing a 21-guage needle and two 20-mL syringes.
  Other Names: Exparel; Multi-Level Intercostal Nerve Block; 0.25% Bupivacaine Hydrochloride; Marcaine
  Arms: Arm 1 "LipoB-I": Liposomal Bupivacaine via Multi-Level Intercostal Nerve Block
Procedure: Arm 2 "LipoB-S": Liposomal Bupivacaine via Serratus Anterior Plane Block — The anesthetic mixture is prepared by combining 266 mg (20 mL) of Liposomal Bupivacaine (Exparel®) with 50 mg (20 mL) of 0.25% Bupivacaine Hydrochloride, creating a mixture of 40 mL. This mixture is administered via serratus anterior plane block.
  One injection is administered by an anesthesiologist in the serratus anterior fascial plane, immediately prior to incision while in the operating room. The total volume of 40 mL is administered using a single-shot technique with a short-bevel, 21-guage needle, ensuring a negative aspiration for blood upon entry, no paresthesia on injection, and incremental injection under ultrasound guidance.
  Other Names: Exparel; Marcaine; Serratus Anterior Plane Block; 0.25% Bupivacaine Hydrochloride
  Arms: Arm 2 "LipoB-S": Liposomal Bupivacaine via Serratus Anterior Plane Block
Procedure: Arm 3 "LipoB-C": Liposomal Bupivacaine Administered via Combination Block — Patients randomized to Arm 3 will receive both a multi-level intercostal nerve block (ICNB) and a serratus anterior plane block (SAPB), with each containing half the dose of Liposomal Bupivacaine (LipoB) as compared to when administered as a single block in Arm 1 and Arm 2. The mixtures are as follows:
  133mg (10mL) LipoB mixed with 25mg (10mL) 0.25% Bupivacaine Hydrochloride and 20mL of saline administered as SAPB by anesthesiologist immediately prior to incision while in the operating room
  AND
  133mg (10mL) LipoB mixed with 25mg (10mL) 0.25% Bupivacaine Hydrochloride and 20mL of saline administered as ICNB prior to closure in at least 5 intercostal spaces as determined by administering surgeon, while in the operating room.
  Other Names: Exparel; Marcaine; 0.25% Bupivacaine Hydrochloride; Combination Block
  Arms: Arm 3 "LipoB-C": Liposomal Bupivacaine via Combination Block

SUMMARY:
The goal of this clinical trial is to assess how the location of local anesthetic medication affects pain control capabilities in adult patients undergoing thoracic(chest)-only minimally invasive surgery. The main questions it aims to answer are:

* Is pain decreased when local analgesia is provided as a combination of serratus anterior plane block and intercostal nerve block when compared to either block administered individually?
* How does location of local analgesia administration impact length-of-stay, cost-of-care, and quality-of-life?

Researchers will compare three treatment options including long-acting local anesthetic (Exparel®) administered as (1) intercostal nerve block, (2) serratus anterior plane block, or (3) combination of intercostal nerve block and serratus anterior plane block to see if pain and opioid use are reduced dependent upon treatment group.

All participants will receive a local anesthetic nerve block. Participants will be asked to describe their pain after surgery and to answer various questionnaires before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Plan to undergo planned (elective) minimally invasive isolated R-VATS procedure, to include pulmonary anatomic resections (anatomic lobectomy, segmentectomy, and wedge resection if performed robotically)
* Age ≥ 18 years old
* Ability to understand and capacity/willingness to sign a written informed consent form

Exclusion Criteria:

* Age < 18 years old
* Unwilling to sign informed consent form, mentally challenged/delayed, or lacking capacity/unable to consent to participation in the trial own their own behalf
* Vulnerable populations
* Incarcerated individuals
* Pregnant individuals
* Breastfeeding individuals
* Individuals with potentially altered pharmacokinetics and metabolism of study drugs
* Renal failure: creatinine ≥ 2, or glomerular filtration rate < 45 mL/min
* Hepatic failure: serum ammonia > 33 mcg/dL and/or Child-Pugh > A
* Individuals suffering from chronic pain
* Individuals taking pre-operative narcotics
* Patients undergoing emergent surgery or urgent surgery for acute, traumatic injuries
* Patients undergoing extra-pleural resections, chest wall resection, pleurectomies, pleurodesis, and decortications
* Planned concurrent abdominal procedure: for example, but not limited to, an esophagectomy
* Patients requiring subcostal transversus abdominis plane (TAP) block
* Use of a rib spreader during thoracic procedure
* Patients admitted to the intensive care unit (ICU) post-operatively while sedated and intubated
* Patients with major post-operative complications
* Wedge resection for pulmonary bleb
* Unanticipated pleurectomy, even if partial
* Surgeon injects superficial wounds with LipoB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
NRS AUC 72 | Post-operative day 0 to post-operative day 3 (if still present in the hospital)
  The investigators will obtain the NRS NRS AUC 72 (units: NRS·hours) (units 0-10) from time 0, entry into the recovery room, to 72 hours after entry into the recovery room. Pain will be assessed by the nursing staff, typically every 4 hours, and by research staff at least once on post-operative days 1-3. The times t0,t1,…,tk in hours within the range of 0 to 72 hours will correspond to NRS scores y0,y1,…,yk. Using the trapezoidal rule over the observed interval (assuming irregular and irregular timing), where: AUC=∑i((yi+yi+1)/2)(ti+1-ti), the maximum NRS·hours would be 10 x 72 hours + 720. If an individual patient measurement is taken off-schedule, the actual time stamps will be utilized. The trapezoidal rule naturally accommodates irregular spacing. If a patient is discharged early, or there is missing data, the AUC will be computed over the observed intervals and reported as time-standardized AUC = (AUC over observed time)/observed hours x 72.
Numeric Rating Scale (NRS) | Post-operative day 0 to post-operative day 3 (if still present in the hospital)
  A pain numeric rating scale will be administered to all patients in the trial from post-operative day 0 to post-operative day 3 in the hospital. Study personnel will gather a NRS value once a day for post-operative day 1-3 and nursing staff will gather a NRS value multiple times a day, typically every 4 hours, per their protocol. Average and maximum values (Likert scale 0-10) will be recorded each day.

SECONDARY OUTCOMES:
Quality-of-Life (Measured by Quality of Recovery Scale) | Post-operative day 1 to post-operative day 3 (if still present in the hospital), as well as at clinic follow-up at 2-5 weeks and via telephone at 90, 180, and 365 days post-operatively
  Investigators will measure post-operative side effects, functional status, and quality-of-life using the Quality of Recovery 15 scale (QR-15). The QR-15 scale measures pain as well as patient daily functioning, enjoyment, relationships, and overall well-being. The QR-15 has previously been validated among the minimally-invasive Thoracic Surgery population, with large-scale studies demonstrating significantly different medial QR-15 scores before to after surgery, with the QR-15 showing significant negative correlations with pain intensity and during coughing in the post-operative period. Further, the pain dimension of the QR-15 correlated to patient "emotional state, physical comfort, and physical independence" at 24, 48, and 72 hours post-operatively. QR-15 may assess nausea, appetite, constipation, and fatigue levels, as well as return to baseline function including return to oral intake, bowel function and ambulation. This scale is favored in clinical use by many anesthesiologists.
Pain Interference via PROMIS Pain Interference (PROMIS-PI) | Clinic follow-up at 2-5 weeks and via telephone at 90, 180, and 365 days post-operatively
  The PROMIS Pain Interference item banks assess self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items probing sleep and enjoyment in life, though the item bank only contains one sleep item. The pain interference short forms are universal rather than disease-specific. All assess pain interference over the past seven days.
Quality of Sleep via PROMIS Sleep Disturbance Short Form (SF) | Post-operative day 1, as well as at clinic follow-up at 2-5 weeks and via telephone at 90, 180, and 365 days post-operatively
  The PROMIS Sleep Disturbance-SF questionnaire will be administered on post-operative day 1, as well as during clinic and telephone follow-up. This questionnaire assesses overall quality of sleep.
Opioid Usage | Post-operative day 0 up to 14 days post-operation
  All opioid usage-including medication type, dosage, and time of administration- will be documented in the medical record. Opioid usage will be converted in a standard fashion to morphine milligram equivalents (MME) per day which will be recorded for all patients. Total cumulative opioid consumption will also be noted. This data will allow the research team to note time until first opioid use after surgery, time until cessation of opioid use after surgery, and whether a patient is utilizing opioids at time of discharge.
Cognitive Function via Neurologic Electrical Response | During surgery (intra-operative EEG) with follow-up assessments (minimal mental state exams) post-operatively up to 14 days post-operation.
  Study subjects will undergo processed electroencephalogram (EEG) monitoring during the procedure. This requires an EEG sensor strip to be placed across the forehead. The use of processed EEG is standard-of-care for anesthesia monitoring during VATS or R-VATS procedures. EEG monitoring intra-operatively will assess neurologic electrical response to treatments (medications, regional nerve blocks, etc.) administered while in the operating room. The anesthesiology team will examine minimal mental state post-operatively per routine care.
Respiratory Function via Incentive Spirometry | Post-operative day 0 up to 14 days post-operation
  An incentive spirometer is a handheld device provided to surgical patients to encourage deep, slow breathing, physiologically re-expanding alveoli that may have collapsed due to under-recruitment during and after surgery. Incentive spirometry maximum volume (mL) is recorded daily as the standard-of-care. Maximum incentive spirometry volume will be noted as a secondary outcome measure as the ability to take deep breaths is often directly correlated to thoracic and chest wall pain.
Adverse Events | Post-operative day 0 to clinic follow-up at 2-5 weeks post-operatively
  All post-operative complications will be documented. All adverse reactions to medications will also be documented. The most common adverse reactions associated with liposomal Bupivacaine are like those of Bupivacaine: nausea, constipation, vomiting, and pyrexia. There have been reports of adverse neurologic reactions with the use of local anesthetics, and toxic blood concentrations depress cardiac conductivity and excitability.
Length of Stay | From date of hospital admission for surgical procedure until date of discharge from hospital, assessed up to 104 weeks.
  Length of hospital stay (days) and length of intensive care unit (ICU) stay will be documented for all patients.
Cost-of-Care | Peri-operative, assessed up to 2 weeks.
  Cost-of-care is an important secondary outcome of this study. The study drugs-Liposomal bupivacaine (Exparel®) and 0.25% bupivacaine hydrochloride (Marcaine®)-are standard of care medications which would be provided to all patients regardless of trial enrollment. The injection volumes of each medication also do not vary between treatment arms. Thus, no difference in cost is incurred for study drugs. Cost-of-care differences arise from equipment costs for ICNB, SAPB, and combination blocks, as well as from billable procedure costs, physician relative value units (RVUs), OR time, and hospital stay time. An activity-based and item-based fee analysis will be performed in combination with LOS and operative time differences between treatment arms to complete a cost analysis as part of this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Inderpal S Sarkaria, MD, MBA, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital at University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Xu HT, Zimmerman J, Bertoch T, Chen L, Chen PJ, Onel E. Efficacy, safety, and pharmacokinetics of CPL-01, an investigational long-acting ropivacaine, in bunionectomy: Results of a phase 2b study. J Foot Ankle Surg. 2025 Mar-Apr;64(2):150-156. doi: 10.1053/j.jfas.2024.09.007. Epub 2024 Sep 19. PMID 39303759
- [Background] Zhang Y, Xian X, Wang F, Zhou B, Wang Y, Wang P, Li Y, Wu Y. Opioid-Free Anesthesia Improved the Quality of Recovery After Thyroidectomy Through Pre-Emptive and Preventive Analgesia: A Randomized Controlled Trial. Drug Des Devel Ther. 2025 Jun 19;19:5243-5254. doi: 10.2147/DDDT.S520856. eCollection 2025. PMID 40552090
- [Background] Xu HT, Zimmerman J, Bertoch T, Chen L, Chen PJ, Onel E. CPL-01, an investigational long-acting ropivacaine, demonstrates safety and efficacy in open inguinal hernia repair. Hernia. 2024 Aug;28(4):1345-1354. doi: 10.1007/s10029-024-03047-3. Epub 2024 May 7. PMID 38713429
- [Background] Administration, U. S. F. a. D. (2022). Statistical Review and Evaluation: P211988Orig1s000StatR. (P211988Orig1s000). U.S. Food and Drug Administration Retrieved from https://www.accessdata.fda.gov/drugsatfda_docs/nda/2022/211988Orig1s000StatR.pdf?utm_source
- [Background] Lang-Illievich K, Wejbora M, Szilagyi IS, Bornemann-Cimenti H. A novel metric for reporting acute postoperative pain correlates more closely with patient satisfaction. Br J Anaesth. 2020 Jun;124(6):e228-e229. doi: 10.1016/j.bja.2020.02.011. Epub 2020 Mar 19. No abstract available. PMID 32199586
- [Background] Viscusi E, Gimbel JS, Pollack RA, Hu J, Lee GC. HTX-011 reduced pain intensity and opioid consumption versus bupivacaine HCl in bunionectomy: phase III results from the randomized EPOCH 1 study. Reg Anesth Pain Med. 2019 May 21:rapm-2019-100531. doi: 10.1136/rapm-2019-100531. Online ahead of print. PMID 31113830
- [Background] Kannampallil T, Galanter WL, Falck S, Gaunt MJ, Gibbons RD, McNutt R, Odwazny R, Schiff G, Vaida AJ, Wilkie DJ, Lambert BL. Characterizing the pain score trajectories of hospitalized adult medical and surgical patients: a retrospective cohort study. Pain. 2016 Dec;157(12):2739-2746. doi: 10.1097/j.pain.0000000000000693. PMID 27548045
- [Background] Ilfeld BM, Malhotra N, Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single-injection peripheral nerve block: a dose-response study. Anesth Analg. 2013 Nov;117(5):1248-56. doi: 10.1213/ANE.0b013e31829cc6ae. PMID 24108252
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Musoro JZ, Coens C, Sprangers MAG, Brandberg Y, Groenvold M, Flechtner HH, Cocks K, Velikova G, Dirven L, Greimel E, Singer S, Pogoda K, Gamper EM, Sodergren SC, Eggermont A, Koller M, Reijneveld JC, Taphoorn MJB, King MT, Bottomley A; EORTC Melanoma, Breast, Head and Neck, Genito-urinary, Gynecological, Gastro-intestinal, Brain, Lung and Quality of Life Groups. Minimally important differences for interpreting EORTC QLQ-C30 change scores over time: A synthesis across 21 clinical trials involving nine different cancer types. Eur J Cancer. 2023 Jul;188:171-182. doi: 10.1016/j.ejca.2023.04.027. Epub 2023 May 7. PMID 37257278
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Davidson EM, Barenholz Y, Cohen R, Haroutiunian S, Kagan L, Ginosar Y. High-dose bupivacaine remotely loaded into multivesicular liposomes demonstrates slow drug release without systemic toxic plasma concentrations after subcutaneous administration in humans. Anesth Analg. 2010 Apr 1;110(4):1018-23. doi: 10.1213/ANE.0b013e3181d26d2a. PMID 20357145
- [Background] Yoon SH, Bae J, Yoon S, Na KJ, Lee HJ. Correlation Between Pain Intensity and Quality of Recovery After Video-Assisted Thoracic Surgery for Lung Cancer Resection. J Pain Res. 2023 Oct 2;16:3343-3352. doi: 10.2147/JPR.S426570. eCollection 2023. PMID 37808464
- [Background] van Dijk JF, van Wijck AJ, Kappen TH, Peelen LM, Kalkman CJ, Schuurmans MJ. The effect of a preoperative educational film on patients' postoperative pain in relation to their request for opioids. Pain Manag Nurs. 2015 Apr;16(2):137-45. doi: 10.1016/j.pmn.2014.05.006. Epub 2014 Sep 22. PMID 25246325
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Background] Grant GJ, Barenholz Y, Bolotin EM, Bansinath M, Turndorf H, Piskoun B, Davidson EM. A novel liposomal bupivacaine formulation to produce ultralong-acting analgesia. Anesthesiology. 2004 Jul;101(1):133-7. doi: 10.1097/00000542-200407000-00021. PMID 15220782
- [Background] Allen MS, Halgren L, Nichols FC 3rd, Cassivi SD, Harmsen WS, Wigle DA, Shen KR, Deschamps C. A randomized controlled trial of bupivacaine through intracostal catheters for pain management after thoracotomy. Ann Thorac Surg. 2009 Sep;88(3):903-10. doi: 10.1016/j.athoracsur.2009.04.139. PMID 19699918
- [Background] Yim AP. Minimizing chest wall trauma in video-assisted thoracic surgery. J Thorac Cardiovasc Surg. 1995 Jun;109(6):1255-6. doi: 10.1016/S0022-5223(95)70217-2. No abstract available. PMID 7776697
- [Background] Bottiger BA, Esper SA, Stafford-Smith M. Pain management strategies for thoracotomy and thoracic pain syndromes. Semin Cardiothorac Vasc Anesth. 2014 Mar;18(1):45-56. doi: 10.1177/1089253213514484. Epub 2013 Dec 12. PMID 24336691
- [Background] Gerdle B, Bjork J, Henriksson C, Bengtsson A. Prevalence of current and chronic pain and their influences upon work and healthcare-seeking: a population study. J Rheumatol. 2004 Jul;31(7):1399-406. PMID 15229963
- [Background] Rogers ML, Duffy JP. Surgical aspects of chronic post-thoracotomy pain. Eur J Cardiothorac Surg. 2000 Dec;18(6):711-6. doi: 10.1016/s1010-7940(00)00569-8. PMID 11113680
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Marcaine TM. https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/018692s015lbl.pdf
- [Background] HIGHLIGHTS of PRESCRIBING INFORMATION. https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/022496s9lbl.pdf
- [Background] Kraft JC, Freeling JP, Wang Z, Ho RJ. Emerging research and clinical development trends of liposome and lipid nanoparticle drug delivery systems. J Pharm Sci. 2014 Jan;103(1):29-52. doi: 10.1002/jps.23773. Epub 2013 Nov 25. PMID 24338748
- [Background] Bulbake U, Doppalapudi S, Kommineni N, Khan W. Liposomal Formulations in Clinical Use: An Updated Review. Pharmaceutics. 2017 Mar 27;9(2):12. doi: 10.3390/pharmaceutics9020012. PMID 28346375
- [Background] Liu P, Chen G, Zhang J. A Review of Liposomes as a Drug Delivery System: Current Status of Approved Products, Regulatory Environments, and Future Perspectives. Molecules. 2022 Feb 17;27(4):1372. doi: 10.3390/molecules27041372. PMID 35209162
- [Background] Research C for DE and. FDA's Efforts to Address the Misuse and Abuse of Opioids. FDA. Published online March 21, 2019. https://www.fda.gov/drugs/information-drug-class/fdas-efforts-address-misuse-and-abuse-opioids
- [Background] National Institute on Drug Abuse. Opioids. National Institute on Drug Abuse. Published 2022. https://nida.nih.gov/research-topics/opioids
- [Background] NCCIH. Chronic Pain and Complementary Health Approaches: Usefulness and Safety. NCCIH. Published January 2023. https://www.nccih.nih.gov/health/chronic-pain-and-complementary-health-approaches-usefulness-and-safety
- [Background] Kianian S, Bansal J, Lee C, Zhang K, Bergese SD. Perioperative multimodal analgesia: a review of efficacy and safety of the treatment options. Anesthesiology and Perioperative Science. 2024;2(1):1-16. doi:https://doi.org/10.1007/s44254-023-00043-1
- [Background] Guerra-Londono CE, Privorotskiy A, Cozowicz C, Hicklen RS, Memtsoudis SG, Mariano ER, Cata JP. Assessment of Intercostal Nerve Block Analgesia for Thoracic Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Nov 1;4(11):e2133394. doi: 10.1001/jamanetworkopen.2021.33394. PMID 34779845
- [Background] Fay K, Patel AD. Should Robot-Assisted Surgery Tolerate or Even Accommodate Less Surgical Dexterity? AMA J Ethics. 2023 Aug 1;25(8):E609-614. doi: 10.1001/amajethics.2023.609. PMID 37535505
- [Background] Julliard W, Krupnick AS. Improving pain after video-assisted thoracoscopic lobectomy-advantages of a wound retractor camera port. J Thorac Dis. 2019 Feb;11(2):341-344. doi: 10.21037/jtd.2018.11.42. No abstract available. PMID 30962968
- [Background] Akter F, Routledge T, Toufektzian L, Attia R. In minor and major thoracic procedures is uniport superior to multiport video-assisted thoracoscopic surgery? Interact Cardiovasc Thorac Surg. 2015 Apr;20(4):550-5. doi: 10.1093/icvts/ivu375. Epub 2015 Jan 28. PMID 25634778
- [Background] McElnay PJ, Molyneux M, Krishnadas R, Batchelor TJ, West D, Casali G. Pain and recovery are comparable after either uniportal or multiport video-assisted thoracoscopic lobectomy: an observation study. Eur J Cardiothorac Surg. 2015 May;47(5):912-5. doi: 10.1093/ejcts/ezu324. Epub 2014 Aug 21. PMID 25147352
- [Background] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Background] Darr C, Cheufou D, Weinreich G, Hachenberg T, Aigner C, Kampe S. Robotic thoracic surgery results in shorter hospital stay and lower postoperative pain compared to open thoracotomy: a matched pairs analysis. Surg Endosc. 2017 Oct;31(10):4126-4130. doi: 10.1007/s00464-017-5464-6. Epub 2017 Mar 8. PMID 28275918
- [Background] Kwon ST, Zhao L, Reddy RM, Chang AC, Orringer MB, Brummett CM, Lin J. Evaluation of acute and chronic pain outcomes after robotic, video-assisted thoracoscopic surgery, or open anatomic pulmonary resection. J Thorac Cardiovasc Surg. 2017 Aug;154(2):652-659.e1. doi: 10.1016/j.jtcvs.2017.02.008. Epub 2017 Feb 14. PMID 28291605
- [Background] Li Z, Liu H, Li L. Video-assisted thoracoscopic surgery versus open lobectomy for stage I lung cancer: A meta-analysis of long-term outcomes. Exp Ther Med. 2012 May;3(5):886-892. doi: 10.3892/etm.2012.485. Epub 2012 Feb 13. PMID 22969988
- [Background] Cerfolio RJ, Price TN, Bryant AS, Sale Bass C, Bartolucci AA. Intracostal sutures decrease the pain of thoracotomy. Ann Thorac Surg. 2003 Aug;76(2):407-11; discussion 411-2. doi: 10.1016/s0003-4975(03)00447-8. PMID 12902074
- [Background] Maguire MF, Latter JA, Mahajan R, Beggs FD, Duffy JP. A study exploring the role of intercostal nerve damage in chronic pain after thoracic surgery. Eur J Cardiothorac Surg. 2006 Jun;29(6):873-9. doi: 10.1016/j.ejcts.2006.03.031. Epub 2006 May 3. PMID 16675262
- [Background] Kaplowitz J, Papadakos PJ. Acute pain management for video-assisted thoracoscopic surgery: an update. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):312-21. doi: 10.1053/j.jvca.2011.04.010. Epub 2011 Jun 25. No abstract available. PMID 21705236
- [Background] Luo F, Cai XJ, Li ZY. Effects of untreated preoperative essential hypertension on post-operative pain after major abdominal surgery. Eur J Pain. 2013 Jan;17(1):94-100. doi: 10.1002/j.1532-2149.2012.00156.x. Epub 2012 Apr 24. PMID 22528813
- [Background] Bruehl S, Chung OY. Interactions between the cardiovascular and pain regulatory systems: an updated review of mechanisms and possible alterations in chronic pain. Neurosci Biobehav Rev. 2004 Jul;28(4):395-414. doi: 10.1016/j.neubiorev.2004.06.004. PMID 15341037
- [Background] Kalkman JC, Visser K, Moen J, Bonsel JG, Grobbee ED, Moons MKG. Preoperative prediction of severe postoperative pain. Pain. 2003 Oct;105(3):415-423. doi: 10.1016/S0304-3959(03)00252-5. PMID 14527702
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Background] Bellville JW, Forrest WH Jr, Miller E, Brown BW Jr. Influence of age on pain relief from analgesics. A study of postoperative patients. JAMA. 1971 Sep 27;217(13):1835-41. No abstract available. PMID 5109724
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Background] Whitlock EL, Diaz-Ramirez LG, Glymour MM, Boscardin WJ, Covinsky KE, Smith AK. Association Between Persistent Pain and Memory Decline and Dementia in a Longitudinal Cohort of Elders. JAMA Intern Med. 2017 Aug 1;177(8):1146-1153. doi: 10.1001/jamainternmed.2017.1622. PMID 28586818
- [Background] Chen WC, Bai YY, Zhang LH, Liu YB, Liu CY, Liang JW, He HF. Prevalence and Predictors of Chronic Postsurgical Pain After Video-Assisted Thoracoscopic Surgery: A Systematic Review and Meta-analysis. Pain Ther. 2023 Feb;12(1):117-139. doi: 10.1007/s40122-022-00439-0. Epub 2022 Oct 13. PMID 36227420
- [Background] Peng Z, Li H, Zhang C, Qian X, Feng Z, Zhu S. A retrospective study of chronic post-surgical pain following thoracic surgery: prevalence, risk factors, incidence of neuropathic component, and impact on qualify of life. PLoS One. 2014 Feb 28;9(2):e90014. doi: 10.1371/journal.pone.0090014. eCollection 2014. PMID 24587187
- [Background] Pedoto A, Noel J, Park BJ, Amar D. Liposomal Bupivacaine Versus Bupivacaine Hydrochloride for Intercostal Nerve Blockade in Minimally Invasive Thoracic Surgery. J Cardiothorac Vasc Anesth. 2021 May;35(5):1393-1398. doi: 10.1053/j.jvca.2020.11.067. Epub 2020 Dec 2. PMID 33376072
- [Background] Marciniak DA, Alfirevic A, Hijazi RM, Ramos DJ, Duncan AE, Gillinov AM, Ahmad U, Murthy SC, Raymond DP. Intercostal Blocks with Liposomal Bupivacaine in Thoracic Surgery: A Retrospective Cohort Study. J Cardiothorac Vasc Anesth. 2021 May;35(5):1404-1409. doi: 10.1053/j.jvca.2020.09.116. Epub 2020 Sep 22. PMID 33067088